CLINICAL TRIAL: NCT05734547
Title: Stepping Together for Children After Trauma: Investigating Effectiveness of a Parent-led, Therapist Assisted Trauma Treatment in Norwegian Municipal Services (The NorStep Study)
Brief Title: Stepping Together for Children After Trauma, Norway
Acronym: NorStep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Center for Violence and Traumatic Stress Studies (Other)
Collaborators: Ministry of Health and Care Services, Norway (Unknown); University of Oslo (Other); King's College London (Other)
Responsible Party: Principal Investigator, Silje Ormhaug, Principal Investigator, Norwegian Center for Violence and Traumatic Stress Studies
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: The NorStep Study
Record Dates: First submitted 2023-02-06; First posted 2023-02-21 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: PTSD; Sleep Disorder; Depressive Symptoms; Quality of Life
Keywords: Posttraumatic stress symptoms; Parent-led treatment; Cost-effectiveness; Childhood trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Wake Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The assessments will be conducted by a clinician from the study group that will be blind to treatment condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stepping Together for Children after Trauma (ST-CT) (Experimental): Parent-led, therapist assisted CBT treatment
  Interventions: Behavioral: Stepping Together for Children after Trauma (ST-CT)
- Usual care (Active Comparator): The types of interventions normally provided in the first-line municipal services
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Stepping Together for Children after Trauma (ST-CT) — ST-CT is Step One of Stepped Care CBT for Children after Trauma (previously called Stepped Care Trauma-focused Cognitive Behavioral Therapy; Salloum et al., 2014). It consists of five components: psychoeducation, stabilization, trauma narrative, in-vivo exposures and consolidation. The parent and child have 11 at-home-meetings and complete tasks in a workbook, Stepping Together (from the Preschool PTSD Treatment by Michael Scheeringa et al), over 6-9 weeks. In addition, there are weekly calls and five sessions with the therapist. Children who meet responder-criteria (i.e., no more than four symptoms of PTSS) continue to a 6-week maintenance phase, after which treatment is complete if the child still meets responder criteria. For those who do not meet responder-criteria, or are not able to complete the workbook, the responsibility for the treatment is transferred from the municipal service level to the corresponding child and adolescent mental health service (BUP).
  Other Names: Part of the treatment previously called Stepped Care Trauma-focused Cognitive Behavioral Therapy
  Arms: Stepping Together for Children after Trauma (ST-CT)
Behavioral: Usual care — Therapists in the control group will provide the treatment they usually provide, and develop a treatment plan in collaboration with the parents. This may consist of individual sessions with the child, parent sessions, group treatment, meetings with the school and other collaborating services, or referral to the second line mental health centres (BUP).
  Arms: Usual care

SUMMARY:
The goal of this randomized controlled trial is to learn about how to effectively help children (aged 7-12) who have developed moderate symptoms of posttraumatic stress after exposure to trauma, and prevent development of more severe problems. The main research questions are:

* Will the parent-led, therapist assisted treatment "Stepping Together for Children after Trauma" (ST-CT) be more effective, compared to usual care, in reducing symptoms of posttraumatic stress, depression and sleep disorders, and in improving daily functioning for children and their parents after trauma?
* Is ST-CT implemented to the municipal first-line services cost-effective?
* Will ST-CT prevent use of health care services and prescribed drugs in the long term?

The children and their non-offending caregivers will be randomized to receive treatment with ST-CT or usual care, and symptoms and general functioning will be assessed at five time-points.

DETAILED DESCRIPTION:
Childhood trauma is a major public health challenge and affects a substantial number of children. Trauma impacts psychological and physical development, as well as long term mental and physical health and behaviour. These adverse outcomes can be prevented through appropriate treatment. Unfortunately, there is a substantial gap between the need for treatment and access to evidence-based care. Low-intensive treatments that utilize and strengthen family resources could contribute to bridging this gap and contribute to improving long-term public health and quality of life.

The Stepped Care Cognitive Behavioral Therapy for Children after Trauma (SC-CBT-CT; Salloum et al. .2014) is a promising intervention for traumatized children that consists of two steps: 1) Stepping Together for Children after Trauma (Stepping Together CT, ST-CT), which is a parent-led, therapist-assisted treatment that takes advantage of and strengthens parent resources; and 2) Trauma-Focused Cognitive Behavioral Therapy (TF-CBT; Cohen et al. 2017) which is a therapist-led treatment provided when Stepping Together CT does not sufficiently help the child. Results from a recent randomized control trial (RCT) conducted in the United States, show that SC-CBT-CT is as effective as standard therapist-led TF-CBT in reducing post-traumatic symptoms, depression, sleep disturbance and parental distress, while simultaneously reducing treatment-related costs by 50% (Salloum et al. 2022). In Norway, a recent pilot study found that the first step, ST-CT, is well accepted by children, parents, and therapists, and is feasible as a first-line intervention in the municipal services (ClinicalTrials.gov Identifier: NCT04073862).

The current study is an RCT with a hybrid effectiveness-implementation design where ST-CT will be implemented to municipal first-line service centers. Participants will be randomized to either the ST-CT or usual care (UC). We will recruit 160 child-parent dyads through 30 participating municipalities from 2023-2025. This will be the first RCT of ST-CT from an independent research group, with the potential for wider implementation which will greatly impact the resources and tools the municipalities have in facing challenges related to childhood trauma.

Aims and data collection:

1) Assess the effectiveness of the parent-led intervention in reducing symptoms on post-traumatic stress, depression, somatic pain and quality of life from both children and caregivers compared to UC. In addition, an objective assessment of quality of sleep will be recorded with a sensor that registers the child's sleep patterns; 2) Evaluate the cost-effectiveness and cost-utility of the ST-CT model; 3) Assess the potential preventive effect of the intervention through long-term follow-up data on use of health services from the Norwegian Patient Registry (NPR), the Norwegian Prescribed Drug Registry (NorPD), and Statistics Norway (SSB); and 4) Investigate barriers and facilitator for implementation, develop culturally adapted treatment material, and an implementation guideline.

Assessments of the children and parents will be conducted by an independent assessor at five time points: T1 = baseline, T2 = after completion of the workbook (ST-CT)/9 weeks (UC); T3 = after the maintenance phase (ST-CT)/ 15 weeks (UC); T4 = 6 months after baseline; T5 = 12 months after baseline.

A secondary aim is to investigate the change-processes within the ST-CT arm, including when during the treatment change in PTSS occurs and how change is related to parenting practices and the child's perceived relationship to their parent.

Assessments related to change-processes will take place in the first 6-9 weeks of treatment, between T1 and T2, for participants in the ST-CT arm only. Specifically, we will collect a short post-traumatic stress symptom assessment (at each parent-child meeting at home, and the first four sessions with the therapist, altogether 15 times), and assess parenting practices and the child's perceived relationship to the parent (the first four sessions with the therapist).

ELIGIBILITY:
Inclusion Criteria:

1. Child is between 7-12 years
2. Exposed to a potentially traumatizing event according to the DSM-5 A-criterion
3. Has a minimum of 5 symptoms of post-traumatic stress (1 symptom must be re-experiencing or avoidance)
4. ≥3 years at the time of the traumatic event to ensure an explicit memory of the event
5. ≥1 month since the traumatic event, according to the diagnostic criteria for PTSD
6. The child must confirm in a conversation alone with the therapist that they feel safe at home and together with the parent and that they are not exposed to ongoing trauma.

Exclusion Criteria:

1. Suspicions of psychosis, active suicidality, serious intellectual disability, or lack of Norwegian skills to complete the workbook
2. A psychotropic medication regime that has not been stable for at least 4 weeks (2 weeks for stimulants/benzodiazepines)
3. Currently receives other trauma treatment.

Caregiver/family exclusion criteria for participation:

1. A caregiver that is the cause of the trauma exposure can neither be the caregiver that leads the treatment nor live in the same household as the child at the time of treatment
2. The caregiver has had a substance use disorder within the past 3 months, suspected suicidality or insufficient Norwegian language skills to complete the workbook/treatment without use of an interpreter.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Child and Adolescent Trauma Screen 2.0 (CATS 2.0) | Baseline (T1)
  The CATS 2.0 assesses child PTSD in the last 4 weeks, according to the DSM-5 and ICD-11 manuals. It includes 15 items of trauma exposure; 20 symptoms of PTS and complex-PTS (intrusions/re-experiencing, avoidance, negative changes in cognition/mood, hyperarousal, and disturbances in self-organization), and 5 items assessing the symptoms' interference on psychosocial functioning. Symptom scores range from 0-60 with higher scores indicating higher levels of PTSD symptoms.
Child and Adolescent Trauma Screen 2.0 (CATS 2.0) | Mid-treatment/ 9 weeks (T2)
  The CATS 2.0 assesses child PTSD in the last 4 weeks, according to the DSM-5 and ICD-11 manuals. It includes 15 items of trauma exposure; 20 symptoms of PTS and complex-PTS (intrusions/re-experiencing, avoidance, negative changes in cognition/mood, hyperarousal, and disturbances in self-organization), and 5 items assessing the symptoms' interference on psychosocial functioning. Symptom scores range from 0-60 with higher scores indicating higher levels of PTSD symptoms.
Child and Adolescent Trauma Screen 2.0 (CATS 2.0) | Post-treatment/ 15 weeks (T3)
  The CATS 2.0 assesses child PTSD in the last 4 weeks, according to the DSM-5 and ICD-11 manuals. It includes 15 items of trauma exposure; 20 symptoms of PTS and complex-PTS (intrusions/re-experiencing, avoidance, negative changes in cognition/mood, hyperarousal, and disturbances in self-organization), and 5 items assessing the symptoms' interference on psychosocial functioning. Symptom scores range from 0-60 with higher scores indicating higher levels of PTSD symptoms.
Child and Adolescent Trauma Screen 2.0 (CATS 2.0) | 6 months follow-up (T4)
  The CATS 2.0 assesses child PTSD in the last 4 weeks, according to the DSM-5 and ICD-11 manuals. It includes 15 items of trauma exposure; 20 symptoms of PTS and complex-PTS (intrusions/re-experiencing, avoidance, negative changes in cognition/mood, hyperarousal, and disturbances in self-organization), and 5 items assessing the symptoms' interference on psychosocial functioning. Symptom scores range from 0-60 with higher scores indicating higher levels of PTSD symptoms.
Child and Adolescent Trauma Screen 2.0 (CATS 2.0) | 12 months follow-up (T5)
  The CATS 2.0 assesses child PTSD in the last 4 weeks, according to the DSM-5 and ICD-11 manuals. It includes 15 items of trauma exposure; 20 symptoms of PTS and complex-PTS (intrusions/re-experiencing, avoidance, negative changes in cognition/mood, hyperarousal, and disturbances in self-organization), and 5 items assessing the symptoms' interference on psychosocial functioning. Symptom scores range from 0-60 with higher scores indicating higher levels of PTSD symptoms.

SECONDARY OUTCOMES:
Short Moods and Feeling Questionnaire (SMFQ) | Baseline (T1)
  The measure has 13 items assessing symptoms of depression during the last 2 weeks. Scores range from 0-26 with higher scores indicating greater depressive symptoms.
Short Moods and Feeling Questionnaire (SMFQ) | Mid-treatment/ 9 weeks (T2)
  The measure has 13 items assessing symptoms of depression during the last 2 weeks. Scores range from 0-26 with higher scores indicating greater depressive symptoms.
Short Moods and Feeling Questionnaire (SMFQ) | Post-treatment/ 15 weeks (T3)
  The measure has 13 items assessing symptoms of depression during the last 2 weeks. Scores range from 0-26 with higher scores indicating greater depressive symptoms.
Short Moods and Feeling Questionnaire (SMFQ) | 6 months follow-up (T4)
  The measure has 13 items assessing symptoms of depression during the last 2 weeks. Scores range from 0-26 with higher scores indicating greater depressive symptoms.
Short Moods and Feeling Questionnaire (SMFQ) | 12 months follow-up (T5)
  The measure has 13 items assessing symptoms of depression during the last 2 weeks. Scores range from 0-26 with higher scores indicating greater depressive symptoms.
Sleep Disturbance Scale for Children (SDSC) | Baseline (T1)
  The scale includes 26 items that covers 6 types of sleep disorders. It is completed by the child's caregiver, and scores range from 26-130, with a higher score indicating more sleep disturbance.
Sleep Disturbance Scale for Children (SDSC) | Mid-treatment/ 9 weeks (T2)
  The scale includes 26 items that covers 6 types of sleep disorders. It is completed by the child's caregiver, and scores range from 26-130, with a higher score indicating more sleep disturbance.
Sleep Disturbance Scale for Children (SDSC) | Post-treatment/ 15 weeks (T3)
  The scale includes 26 items that covers 6 types of sleep disorders. It is completed by the child's caregiver, and scores range from 26-130, with a higher score indicating more sleep disturbance.
Sleep Disturbance Scale for Children (SDSC) | 6 months follow-up (T4)
  The scale includes 26 items that covers 6 types of sleep disorders. It is completed by the child's caregiver, and scores range from 26-130, with a higher score indicating more sleep disturbance.
Sleep Disturbance Scale for Children (SDSC) | 12 months follow-up (T5)
  The scale includes 26 items that covers 6 types of sleep disorders. It is completed by the child's caregiver, and scores range from 26-130, with a higher score indicating more sleep disturbance.
Children's Post-Traumatic Cognitions Inventory Short (CPTCI-S) | Baseline (T1)
  The scale includes 10 items covering the two components "Disturbing and permanent change" and "Feeble person in a scary world". Scores range from 10-40, with higher scores indicating greater post-traumatic cognitions.
Children's Post-Traumatic Cognitions Inventory Short (CPTCI-S) | Mid-treatment/ 9 weeks (T2)
  The scale includes 10 items covering the two components "Disturbing and permanent change" and "Feeble person in a scary world". Scores range from 10-40, with higher scores indicating greater post-traumatic cognitions.
Children's Post-Traumatic Cognitions Inventory Short (CPTCI-S) | Post-treatment/ 15 weeks (T3)
  The scale includes 10 items covering the two components "Disturbing and permanent change" and "Feeble person in a scary world". Scores range from 10-40, with higher scores indicating greater post-traumatic cognitions.
Children's Post-Traumatic Cognitions Inventory Short (CPTCI-S) | 6 months follow-up (T4)
  The scale includes 10 items covering the two components "Disturbing and permanent change" and "Feeble person in a scary world". Scores range from 10-40, with higher scores indicating greater post-traumatic cognitions.
Children's Post-Traumatic Cognitions Inventory Short (CPTCI-S) | 12 months follow-up (T5)
  The scale includes 10 items covering the two components "Disturbing and permanent change" and "Feeble person in a scary world". Scores range from 10-40, with higher scores indicating greater post-traumatic cognitions.
The Parent Child Communication Scale, child version (PCCSc) | Baseline (T1)
  10 items covering the child's perception of their communication with their parents. Scores range from 0-40, with higher scores indicating better communication with the parent.
The Parent Child Communication Scale, child version (PCCSc) | Mid-treatment/ 9 weeks (T2)
  10 items covering the child's perception of their communication with their parents. Scores range from 0-40, with higher scores indicating better communication with the parent.
The Parent Child Communication Scale, child version (PCCSc) | Post-treatment/ 15 weeks (T3)
  10 items covering the child's perception of their communication with their parents. Scores range from 0-40, with higher scores indicating better communication with the parent.
The Parent Child Communication Scale, child version (PCCSc) | 6 months follow-up (T4)
  10 items covering the child's perception of their communication with their parents. Scores range from 0-40, with higher scores indicating better communication with the parent.
The Parent Child Communication Scale, child version (PCCSc) | 12 months follow-up (T5)
  10 items covering the child's perception of their communication with their parents. Scores range from 0-40, with higher scores indicating better communication with the parent.
Kidscreen 52 - The Parent Relations and Home Life dimension | Baseline (T1)
  The scale has 6 items covering the child's perceptions of being loved, understood, and being able to talk to their parents, during the last week. Scores range from 6-30, with higher scores indicating better relationships and home-life.
Kidscreen 52 - The Parent Relations and Home Life dimension | Mid-treatment/ 9 weeks (T2)
  The scale has 6 items covering the child's perceptions of being loved, understood, and being able to talk to their parents, during the last week. Scores range from 6-30, with higher scores indicating better relationships and home-life.
Kidscreen 52 - The Parent Relations and Home Life dimension | Post-treatment/ 15 weeks (T3)
  The scale has 6 items covering the child's perceptions of being loved, understood, and being able to talk to their parents, during the last week. Scores range from 6-30, with higher scores indicating better relationships and home-life.
Kidscreen 52 - The Parent Relations and Home Life dimension | 6 months follow-up (T4)
  The scale has 6 items covering the child's perceptions of being loved, understood, and being able to talk to their parents, during the last week. Scores range from 6-30, with higher scores indicating better relationships and home-life.
Kidscreen 52 - The Parent Relations and Home Life dimension | 12 months follow-up (T5)
  The scale has 6 items covering the child's perceptions of being loved, understood, and being able to talk to their parents, during the last week. Scores range from 6-30, with higher scores indicating better relationships and home-life.
Kidscreen 52 - The Parent Relations and Home Life dimension | Every 2 weeks between T1 and T2 (3 times)
  The scale has 6 items covering the child's perceptions of being loved, understood, and being able to talk to their parents, during the last week. Scores range from 6-30, with higher scores indicating better relationships and home-life. For the children in the ST-CT arm only, we include these additional measuring points of Parent Relations to be able to explore change-processed during treatment with ST-CT (assessment at the first four sessions with the therapist).
Strengths and Difficulties Questionnaire (SDQ) - Parent and Teacher report | Baseline (T1)
  The SDQ includes 25 items covering five areas of clinical interest: hyperactivity/inattention, emotional symptoms, conduct problems, peer relation problems, and prosocial behaviors. The four first areas (20 items) can be summed to give an overall picture of difficulties, with scores ranging from 0-40, or kept as two subscales (internalizing and externalizing) of 10 items each. Higher scores indicate more difficulties. The fifth area, prosocial behavior, is kept as a separate scale from 0-10 where a higher score indicates more prosocial behaviors/strengths.
Strengths and Difficulties Questionnaire (SDQ) - Parent and Teacher report | Mid-treatment/ 9 weeks (T2)
  The SDQ includes 25 items covering five areas of clinical interest: hyperactivity/inattention, emotional symptoms, conduct problems, peer relation problems, and prosocial behaviors. The four first areas (20 items) can be summed to give an overall picture of difficulties, with scores ranging from 0-40, or kept as two subscales (internalizing and externalizing) of 10 items each. Higher scores indicate more difficulties. The fifth area, prosocial behavior, is kept as a separate scale from 0-10 where a higher score indicates more prosocial behaviors/strengths.
Strengths and Difficulties Questionnaire (SDQ) - Parent and Teacher report | Post-treatment/ 15 weeks (T3)
  The SDQ includes 25 items covering five areas of clinical interest: hyperactivity/inattention, emotional symptoms, conduct problems, peer relation problems, and prosocial behaviors. The four first areas (20 items) can be summed to give an overall picture of difficulties, with scores ranging from 0-40, or kept as two subscales (internalizing and externalizing) of 10 items each. Higher scores indicate more difficulties. The fifth area, prosocial behavior, is kept as a separate scale from 0-10 where a higher score indicates more prosocial behaviors/strengths.
Strengths and Difficulties Questionnaire (SDQ) - Parent and Teacher report | 6 months follow-up (T4)
  The SDQ includes 25 items covering five areas of clinical interest: hyperactivity/inattention, emotional symptoms, conduct problems, peer relation problems, and prosocial behaviors. The four first areas (20 items) can be summed to give an overall picture of difficulties, with scores ranging from 0-40, or kept as two subscales (internalizing and externalizing) of 10 items each. Higher scores indicate more difficulties. The fifth area, prosocial behavior, is kept as a separate scale from 0-10 where a higher score indicates more prosocial behaviors/strengths.
Strengths and Difficulties Questionnaire (SDQ) - Parent and Teacher report | 12 months follow-up (T5)
  The SDQ includes 25 items covering five areas of clinical interest: hyperactivity/inattention, emotional symptoms, conduct problems, peer relation problems, and prosocial behaviors. The four first areas (20 items) can be summed to give an overall picture of difficulties, with scores ranging from 0-40, or kept as two subscales (internalizing and externalizing) of 10 items each. Higher scores indicate more difficulties. The fifth area, prosocial behavior, is kept as a separate scale from 0-10 where a higher score indicates more prosocial behaviors/strengths.
Child Health Utility instrument (CHU9D) | Baseline (T1)
  The CHU9D is a measure of health-related quality of life (HRQoL). The scale covers 9 dimensions such as feeling worried, tired, annoyed, and not being able to complete school-work, daily activities and chores. Each dimension has 5 response levels, and higher scores indicate lower HRQoL.
Child Health Utility instrument (CHU9D) | Mid-treatment/ 9 weeks (T2)
  The CHU9D is a measure of health-related quality of life (HRQoL). The scale covers 9 dimensions such as feeling worried, tired, annoyed, and not being able to complete school-work, daily activities and chores. Each dimension has 5 response levels, and higher scores indicate lower HRQoL.
Child Health Utility instrument (CHU9D) | Post-treatment/ 15 weeks (T3)
  The CHU9D is a measure of health-related quality of life (HRQoL). The scale covers 9 dimensions such as feeling worried, tired, annoyed, and not being able to complete school-work, daily activities and chores. Each dimension has 5 response levels, and higher scores indicate lower HRQoL.
Child Health Utility instrument (CHU9D) | 6 months follow-up (T4)
  The CHU9D is a measure of health-related quality of life (HRQoL). The scale covers 9 dimensions such as feeling worried, tired, annoyed, and not being able to complete school-work, daily activities and chores. Each dimension has 5 response levels, and higher scores indicate lower HRQoL.
Child Health Utility instrument (CHU9D) | 12 months follow-up (T5)
  The CHU9D is a measure of health-related quality of life (HRQoL). The scale covers 9 dimensions such as feeling worried, tired, annoyed, and not being able to complete school-work, daily activities and chores. Each dimension has 5 response levels, and higher scores indicate lower HRQoL.
Kidscreen 27: Friends and school dimensions | Baseline (T1)
  The scales consists of 4 questions regarding the child's relationship to their friends, and 4 items regarding school functioning during the last week. Items are scored on a 5-point scale, ranging from 4-20 for each subscale. Higher scores indicate better functioning.
Kidscreen 27: Friends and School dimension | Mid-treatment/9 weeks (T2)
  The scales consists of 4 questions regarding the child's relationship to their friends, and 4 items regarding school functioning during the last week. Items are scored on a 5-point scale, ranging from 4-20 for each subscale. Higher scores indicate better functioning.
Kidscreen 27: Friends and School dimension | Post-treatment/15 weeks (T3)
  The scales consists of 4 questions regarding the child's relationship to their friends, and 4 items regarding school functioning during the last week. Items are scored on a 5-point scale, ranging from 4-20 for each subscale. Higher scores indicate better functioning.
Kidscreen 27: Friends and School dimension | 6 months follow-up (T4)
  The scales consists of 4 questions regarding the child's relationship to their friends, and 4 items regarding school functioning during the last week. Items are scored on a 5-point scale, ranging from 4-20 for each subscale. Higher scores indicate better functioning.
Kidscreen 27: Friends and School dimension | 12 months follow-up (T5)
  The scales consists of 4 questions regarding the child's relationship to their friends, and 4 items regarding school functioning during the last week. Items are scored on a 5-point scale, ranging from 4-20 for each subscale. Higher scores indicate better functioning.
Children's somatic symptoms inventory short form (CSSI-8) | Baseline (T1)
  The scale consists of 8 items covering pain and somatic symptoms during the last 2 weeks. Scores range from 0-32 with higher scores indicating more somatic symptoms.
Children's somatic symptoms inventory short form (CSSI-8) | Mid-treatment/ 9 weeks (T2)
  The scale consists of 8 items covering pain and somatic symptoms during the last 2 weeks. Scores range from 0-32 with higher scores indicating more somatic symptoms.
Children's somatic symptoms inventory short form (CSSI-8) | Post-treatment/ 15 weeks (T3)
  The scale consists of 8 items covering pain and somatic symptoms during the last 2 weeks. Scores range from 0-32 with higher scores indicating more somatic symptoms.
Children's somatic symptoms inventory short form (CSSI-8) | 6 months follow-up (T4)
  The scale consists of 8 items covering pain and somatic symptoms during the last 2 weeks. Scores range from 0-32 with higher scores indicating more somatic symptoms.
Children's somatic symptoms inventory short form (CSSI-8) | 12 months follow-up (T5)
  The scale consists of 8 items covering pain and somatic symptoms during the last 2 weeks. Scores range from 0-32 with higher scores indicating more somatic symptoms.
Child sleep quality: objective measure and sleep diary | 7 days before treatment starts
  A non-contact sensor (Somnofy radar, Vital Things A/S) will be used to assess the child's sleep quality in 7 days before treatment start. The sensor registers the child's movement, respiration frequency and sleep quality during the night. A sleep diary will be completed for the same 7 days, with parents recording: when their child falls asleep, wakes up, time taken to fall asleep, awake periods during the night and how well they slept; and the child reporting: if they woke up at time, how many times and how well they slept.
Child sleep quality: objective measure and sleep diary | 7 days post-treatment/ after 15 weeks
  A non-contact sensor (Somnofy radar, Vital Things A/S) will be used to assess the child's sleep quality in 7 days before treatment start. The sensor registers the child's movement, respiration frequency and sleep quality during the night. A sleep diary will be completed for the same 7 days, with parents recording: when their child falls asleep, wakes up, time taken to fall asleep, awake periods during the night and how well they slept; and the child reporting: if they woke up at time, how many times and how well they slept.
The Rage Outburst and Anger Rating Scale (ROARS) | Baseline (T1)
  3 items where the parent rates the frequency, intensity and duration of the child's anger outbursts in the last 7 days. Each item is scored on a 4-point scale, and the sum score ranges from 0 to 9, with a higher score indicating more severe anger outbursts.
The Rage Outburst and Anger Rating Scale (ROARS) | Mid-treatment/9 weeks (T2)
  3 items where the parent rates the frequency, intensity and duration of the child's anger outbursts in the last 7 days. Each item is scored on a 4-point scale, and the sum score ranges from 0 to 9, with a higher score indicating more severe anger outbursts.
The Rage Outburst and Anger Rating Scale (ROARS) | Post-treatment/15 weeks (T3)
  3 items where the parent rates the frequency, intensity and duration of the child's anger outbursts in the last 7 days. Each item is scored on a 4-point scale, and the sum score ranges from 0 to 9, with a higher score indicating more severe anger outbursts.
The Rage Outburst and Anger Rating Scale (ROARS) | 6 months follow-up (T4)
  3 items where the parent rates the frequency, intensity and duration of the child's anger outbursts in the last 7 days. Each item is scored on a 4-point scale, and the sum score ranges from 0 to 9, with a higher score indicating more severe anger outbursts.
The Rage Outburst and Anger Rating Scale (ROARS) | 12 months follow-up (T5)
  3 items where the parent rates the frequency, intensity and duration of the child's anger outbursts in the last 7 days. Each item is scored on a 4-point scale, and the sum score ranges from 0 to 9, with a higher score indicating more severe anger outbursts.
The Child and Adolescent Serive Use Schedule (CA-SUS) | Baseline (T1)
  The parents report the total amount of health and social care services the child has received, including type of services and quantity, and the parents' days of absence from work. The type of services, quantity and parents' work-absence will be transformed to reflect costs related to services used, using cost units from the corresponding financial years.
  At baseline, service use in the last 6 months will be recorded.
The Child and Adolescent Serive Use Schedule (CA-SUS) | Mid-treatment/9 weeks (T2)
  The parents report the total amount of health and social care services the child has received, including type of services and quantity, and the parents' days of absence from work. The type of services, quantity and parents' work-absence will be transformed to reflect costs related to services used, using cost units from the corresponding financial years.
  At T2, service use in the period since T1 will be recorded.
The Child and Adolescent Serive Use Schedule (CA-SUS) | Post-treatment/15 weeks (T3)
  The parents report the total amount of health and social care services the child has received, including type of services and quantity, and the parents' days of absence from work. The type of services, quantity and parents' work-absence will be transformed to reflect costs related to services used, using cost units from the corresponding financial years.
  At T3, service use in the period since T2 will be recorded.
The Child and Adolescent Serive Use Schedule (CA-SUS) | 6 months follow-up (T4)
  The parents report the total amount of health and social care services the child has received, including type of services and quantity, and the parents' days of absence from work. The type of services, quantity and parents' work-absence will be transformed to reflect costs related to services used, using cost units from the corresponding financial years.
  At T4, service use in the period since T3 will be recorded.
The Child and Adolescent Serive Use Schedule (CA-SUS) | 12 months follow-up (T5)
  The parents report the total amount of health and social care services the child has received, including type of services and quantity, and the parents' days of absence from work. The type of services, quantity and parents' work-absence will be transformed to reflect costs related to services used, using cost units from the corresponding financial years.
  At T5, service use in the period since T4 will be recorded.
The ICD-11 criteria of the Child and Adolescent Trauma Screen 2.0 (CATS 2.0) | Twice a week between T1 and T2 (at the at-home meetings, 15 assessments)
  We will use the 9 items that are prerequisites for assessing both an ICD-11 PTSD diagnosis (complex and non-complex) and and DSM-5 diagnosis, in the CATS 2.0 to assess change processes for the children in the ST-CT arm only. This will be assessed up to 15 times in the period between T1 and T2 (at 11 home parent-child meetings and 4 therapist sessions).

OTHER OUTCOMES:
Stressful Life-Events Screening Questionnaire (SLESQ) | Baseline (T1)
  SLESQ assesses the parent's life-time exposure to 15 potentially traumatizing events, with scores ranging from 0-15.
Stressful Life-Events Screening Questionnaire (SLESQ) | Mid-treatment/ 9 weeks (T2)
  SLESQ assesses the parent's exposure to 15 potentially traumatizing events since the last assessment. Scores range from 0-15.
Stressful Life-Events Screening Questionnaire (SLESQ) | Post-treatment/ 15 weeks (T3)
  SLESQ assesses the parent's exposure to 15 potentially traumatizing events since the last assessment. Scores range from 0-15.
Stressful Life-Events Screening Questionnaire (SLESQ) | 6 months follow-up (T4)
  SLESQ assesses the parent's exposure to 15 potentially traumatizing events since the last assessment. Scores range from 0-15.
Stressful Life-Events Screening Questionnaire (SLESQ) | 12 months follow-up (T5)
  SLESQ assesses the parent's exposure to 15 potentially traumatizing events since the last assessment. Scores range from 0-15.
International Trauma Questionnaire (ITQ) | Baseline (T1)
  The ITQ assesses symptoms of post-traumatic stress disorder (PTSD) and Complex PTSD according to the ICD-11. It includes 18 items, and scores range from 0-90, with higher scores indicating greater PTSD
International Trauma Questionnaire (ITQ) | Mid-treatment/ 9 weeks (T2)
  The ITQ assesses symptoms of post-traumatic stress disorder (PTSD) and Complex PTSD according to the ICD-11. It includes 18 items, and scores range from 0-90, with higher scores indicating greater PTSD
International Trauma Questionnaire (ITQ) | Post-treatment/ 15 weeks (T3)
  The ITQ assesses symptoms of post-traumatic stress disorder (PTSD) and Complex PTSD according to the ICD-11. It includes 18 items, and scores range from 0-90, with higher scores indicating greater PTSD
International Trauma Questionnaire (ITQ) | 6 months follow-up (T4)
  The ITQ assesses symptoms of post-traumatic stress disorder (PTSD) and Complex PTSD according to the ICD-11. It includes 18 items, and scores range from 0-90, with higher scores indicating greater PTSD
International Trauma Questionnaire (ITQ) | 12 months follow-up (T5)
  The ITQ assesses symptoms of post-traumatic stress disorder (PTSD) and Complex PTSD according to the ICD-11. It includes 18 items, and scores range from 0-90, with higher scores indicating greater PTSD
Hopkins Symptom Check List 25 (HSCL-25) | Baseline (T1)
  The HSCL-25 measures the parent's symptoms of anxiety and depression during the last 2 weeks. Scores range from 25-100, with higher scores indicating greater anxiety and depression.
Hopkins Symptom Check List 25 (HSCL-25) | Mid-treatment/ 9 weeks (T2)
  The HSCL-25 measures the parent's symptoms of anxiety and depression during the last 2 weeks. Scores range from 25-100, with higher scores indicating greater anxiety and depression.
Hopkins Symptom Check List 25 (HSCL-25) | Post-treatment/ 15 weeks (T3)
  The HSCL-25 measures the parent's symptoms of anxiety and depression during the last 2 weeks. Scores range from 25-100, with higher scores indicating greater anxiety and depression.
Hopkins Symptom Check List 25 (HSCL-25) | 6 months follow-up (T4)
  The HSCL-25 measures the parent's symptoms of anxiety and depression during the last 2 weeks. Scores range from 25-100, with higher scores indicating greater anxiety and depression.
Hopkins Symptom Check List 25 (HSCL-25) | 12 months follow-up (T5)
  The HSCL-25 measures the parent's symptoms of anxiety and depression during the last 2 weeks. Scores range from 25-100, with higher scores indicating greater anxiety and depression.
Parents Emotional Reactions Questionnaire (PERQ) | Baseline (T1)
  The scale consists of 15 items covering the parent's emotional reactions (distress, shame and guilt) to their child's trauma during the last 2 weeks. In this study, item 15 (have you felt guilty about not discovering your child's trauma sooner) will not be included, as it is not relevant for many participants. Scores will range from 14-70 with higher scores indicating greater emotional reactions.
Parents Emotional Reactions Questionnaire (PERQ) | Mid-treatment/ 9 weeks (T2)
  The scale consists of 15 items covering the parent's emotional reactions (distress, shame and guilt) to their child's trauma during the last 2 weeks. In this study, item 15 (have you felt guilty about not discovering your child's trauma sooner) will not be included, as it is not relevant for many participants. Scores will range from 14-70 with higher scores indicating greater emotional reactions.
Parents Emotional Reactions Questionnaire (PERQ) | Post-treatment/ 15 weeks (T3)
  The scale consists of 15 items covering the parent's emotional reactions (distress, shame and guilt) to their child's trauma during the last 2 weeks. In this study, item 15 (have you felt guilty about not discovering your child's trauma sooner) will not be included, as it is not relevant for many participants. Scores will range from 14-70 with higher scores indicating greater emotional reactions.
Parents Emotional Reactions Questionnaire (PERQ) | 6 months follow-up (T4)
  The scale consists of 15 items covering the parent's emotional reactions (distress, shame and guilt) to their child's trauma during the last 2 weeks. In this study, item 15 (have you felt guilty about not discovering your child's trauma sooner) will not be included, as it is not relevant for many participants. Scores will range from 14-70 with higher scores indicating greater emotional reactions.
Parents Emotional Reactions Questionnaire (PERQ) | 12 months follow-up (T5)
  The scale consists of 15 items covering the parent's emotional reactions (distress, shame and guilt) to their child's trauma during the last 2 weeks. In this study, item 15 (have you felt guilty about not discovering your child's trauma sooner) will not be included, as it is not relevant for many participants. Scores will range from 14-70 with higher scores indicating greater emotional reactions.
Parent Trauma Response Questionnaire (PTRQ), Child coping dimension | Baseline (T1)
  The scale consists of 20 items covering five different types of parent strategies: behavioral avoidance, cognitive avoidance, overprotection, maintaining pre-trauma routines, and approach coping. Scores range from 0-80, with higher scores indicating more of the parent strategy.
Parent Trauma Response Questionnaire (PTRQ), Child coping dimension | Mid-treatment/ 9 weeks (T2)
  The scale consists of 20 items covering five different types of parent strategies: behavioral avoidance, cognitive avoidance, overprotection, maintaining pre-trauma routines, and approach coping. Scores range from 0-80, with higher scores indicating more of the parent strategy.
Parent Trauma Response Questionnaire (PTRQ), Child coping dimension | Post-treatment/ 15 weeks (T3)
  The scale consists of 20 items covering five different types of parent strategies: behavioral avoidance, cognitive avoidance, overprotection, maintaining pre-trauma routines, and approach coping. Scores range from 0-80, with higher scores indicating more of the parent strategy.
Parent Trauma Response Questionnaire (PTRQ), Child coping dimension | 6 months follow-up (T4)
  The scale consists of 20 items covering five different types of parent strategies: behavioral avoidance, cognitive avoidance, overprotection, maintaining pre-trauma routines, and approach coping. Scores range from 0-80, with higher scores indicating more of the parent strategy.
Parent Trauma Response Questionnaire (PTRQ), Child coping dimension | 12 months follow-up (T5)
  The scale consists of 20 items covering five different types of parent strategies: behavioral avoidance, cognitive avoidance, overprotection, maintaining pre-trauma routines, and approach coping. Scores range from 0-80, with higher scores indicating more of the parent strategy.
Implementation Leadership Scale (ILS) | Before training
  The scale consists of 12 items covering proactive, knowledgeable, supportive and perseverant leadership, and will be completed by the participating therapists. Scores range from 0-48, with higher scores indicating greater implementation leadership.
Implementation Leadership Scale (ILS) | 4 months after training
  The scale consists of 12 items covering proactive, knowledgeable, supportive and perseverant leadership, and will be completed by the participating therapists. Scores range from 0-48, with higher scores indicating greater implementation leadership.
Implementation Leadership Scale (ILS) | 8 months after training
  The scale consists of 12 items covering proactive, knowledgeable, supportive and perseverant leadership, and will be completed by the participating therapists. Scores range from 0-48, with higher scores indicating greater implementation leadership.
Implementation Leadership Scale (ILS) | 12 months after training
  The scale consists of 12 items covering proactive, knowledgeable, supportive and perseverant leadership, and will be completed by the participating therapists. Scores range from 0-48, with higher scores indicating greater implementation leadership.
Professional Quality of Life Scale (ProQOL-V) | Before training
  The ProQOL consists of 30 items assessing compassion satisfaction, burnout and secondary traumatic stress in therapists. Scores range from 30-150, with higher scores indicating higher satisfaction/ burnout/ secondary traumatic stress.
Professional Quality of Life Scale (ProQOL-V) | 4 months after training
  The ProQOL consists of 30 items assessing compassion satisfaction, burnout and secondary traumatic stress in therapists. Scores range from 30-150, with higher scores indicating higher satisfaction/ burnout/ secondary traumatic stress.
Professional Quality of Life Scale (ProQOL-V) | 8 months after training
  The ProQOL consists of 30 items assessing compassion satisfaction, burnout and secondary traumatic stress in therapists. Scores range from 30-150, with higher scores indicating higher satisfaction/ burnout/ secondary traumatic stress.
Professional Quality of Life Scale (ProQOL-V) | 12 months after training
  The ProQOL consists of 30 items assessing compassion satisfaction, burnout and secondary traumatic stress in therapists. Scores range from 30-150, with higher scores indicating higher satisfaction/ burnout/ secondary traumatic stress.
Turnover Intention Scale (TIS) | Before training
  The TIS includes 6 items measuring therapist's turnover intention. Scores range from 6-30 with higher scores indicating greater turnover intentions.
Turnover Intention Scale (TIS) | 4 months after training
  The TIS includes 6 items measuring therapist's turnover intention. Scores range from 6-30 with higher scores indicating greater turnover intentions.
Turnover Intention Scale (TIS) | 8 months after training
  The TIS includes 6 items measuring therapist's turnover intention. Scores range from 6-30 with higher scores indicating greater turnover intentions.
Turnover Intention Scale (TIS) | 12 months after training
  The TIS includes 6 items measuring therapist's turnover intention. Scores range from 6-30 with higher scores indicating greater turnover intentions.

CONTACTS AND LOCATIONS:
Overall Officials: Silje M Ormhaug, Principal Investigator — Norwegian Center for Violence and Traumatic Stress Studies (NKVTS)
Locations (2):
- Norway (2):
  - Asker kommune, Asker
  - NKVTS, Oslo

IPD SHARING:
Plan to Share IPD: Yes
De-coded individual participant data will be made available after data inclusion upon participants' written consent.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2026-2032
Access Criteria: Receiving party must follow the general data protection pegulation (GDPR).

REFERENCES:
- [Background] Salloum A, Lu Y, Chen H, Quast T, Cohen JA, Scheeringa MS, Salomon K, Storch EA. Stepped Care Versus Standard Care for Children After Trauma: A Randomized Non-Inferiority Clinical Trial. J Am Acad Child Adolesc Psychiatry. 2022 Aug;61(8):1010-1022.e4. doi: 10.1016/j.jaac.2021.12.013. Epub 2022 Jan 12. PMID 35032578
- [Background] Salloum A, Scheeringa MS, Cohen JA, Storch EA. Development of Stepped Care Trauma-Focused Cognitive-Behavioral Therapy for Young Children. Cogn Behav Pract. 2014 Feb 1;21(1):97-108. doi: 10.1016/j.cbpra.2013.07.004. PMID 25411544
- [Background] Cohen JA, Mannarino AP, Deblinger E. Treating Trauma and Traumatic Grief in Children and Adolescents. 2nd ed. New York: Guilford Press; 2017
- [Derived] Ormhaug SM, Jensen TK, Porcheret KL, Andreassen AL, Byford S, Fagermoen EMK, Gurandsrud P, Haabrekke KJO, Lindebo Knutsen M, Paivarinne HM, Skjaervo I. Stepping together for children after trauma: protocol for a randomized controlled trial of a parent-led treatment in first-line services (NorStep Study). Eur J Psychotraumatol. 2025 Dec;16(1):2555047. doi: 10.1080/20008066.2025.2555047. Epub 2025 Sep 17. PMID 40958761